CLINICAL TRIAL: NCT06412965
Title: Evaluation of the Reliability of Effect of Rimegepant for the Acute Treatment of Migraine Across Multiple Attacks
Brief Title: Reliability of Rimegepant or Triptans for the Acute Treatment of Migraine
Acronym: Adelphi DSP
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C4951066
Record Dates: First submitted 2024-04-16; First posted 2024-05-14 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-11

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Rimegepant: Cohort of patients treated with rimegepant
- Triptans: Cohort of patients treated with triptans

SUMMARY:
This protocol describes the analysis of the Adelphi Real World (ARW) Migraine Disease Specific Programme(TM) 2022, a cross-sectional study which used both physician and patient surveys to assess the perception of the acute treatment for migraine attacks.

DETAILED DESCRIPTION:
This is a retrospective database study that aims to explore the reliability of effect with acute use of Rimegepant or triptans, to evaluate the satisfaction with Rimegepant or triptans, to evaluate willingness to continue using Rimegepant or triptans, and to explore proportion optimized on treatment with Rimegepant or triptans. The data will be extracted from the Adelphi Real World (ARW) Migraine Disease Specific ProgrammeTM (DSP) 2022 database, which was conducted across a number of countries including United States, between May 2022 and November 2022. The DSP was an observational study of clinical practice. Treatment practice data were collected by physicians (physician survey) who were asked to provide information for the next 10 patients consulting for migraine. These patients were then invited to fill out a self-completion form (patient survey) providing their own assessment on the disease and treatments.

ELIGIBILITY:
Inclusion criteria

* Patients who have episodic and/or chronic migraine
* Patients age > 18
* Currently prescribed rimegepant OR triptans for the acute treatment of migraine

Exclusion criteria

* currently prescribed rimegepant for prevention of migraine or for both the acute treatment & prevention of migraine
* Rimegepant group: currently prescribed an acute treatment for migraine and other than rimegepant
* Triptan Group: currently prescribed an acute treatment for migraine other than triptans

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Physician personally responsible for treatment decision of migraine patients were enrolled in the survey. Each physician then enrolled consecutive patients to complete a patient self-completion questionnaire.
Sampling Method: Non-Probability Sample
Enrollment: 528 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-01-03 (Actual); Study Completion 2024-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4951066

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data was extracted from Adelphi Real World (ARW) Migraine VII Disease Specific Programme (DSP) 2022 database. Participants diagnosed with migraine and prescribed rimegepant or triptans as an acute treatment for their migraine in the US, were recruited into the Migraine VII DSP US between May 2022 and November 2022. This retrospective observational study comprised secondary data analysis of DSP data.
Groups:
- Rimegepant: Participants who in a real world setting under routine clinical practice were prescribed rimegepant for the acute treatment of migraine and their data was observed retrospectively in this study.
- Triptans: Participants who in a real world setting under routine clinical practice were prescribed triptans for the acute treatment of migraine and their data was observed retrospectively in this study.
Period: Overall Study
Arm/Group | Rimegepant | Triptans
Started | 91 | 437
Completed | 91 | 437
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all participants who met eligibility criteria and whose data was retrospectively observed in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rimegepant | Triptans | Total
Number analyzed (Participants) | 91 | 437 | 528
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.01 (13.11) | 38.98 (13.4) | 38.99 (13.34)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Number Analyzed = Number of participants who were evaluable and had non-missing values.
  Participants
    number analyzed (Participants) | 89 | 437 | 526
    Female | 66 | 309 | 375
    Male | 23 | 128 | 151
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Some participants recorded as more than one ethnicity, hence the total for all categories is higher than the total number analyzed.
  Participants
    White/Caucasian | 65 | 304 | 369
    African American | 12 | 65 | 77
    Native American | 1 | 1 | 2
    Asian (Indian subcontinent) | 0 | 8 | 8
    South-East Asian | 1 | 8 | 9
    Asian (other) | 2 | 8 | 10
    Hispanic / Latino / Latina | 8 | 38 | 46
    Middle Eastern | 2 | 8 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Failed to Achieve Pain Freedom Within 2 Hours Post Dose (Physician Perspective)
Description: Physicians responded as "Yes" or "No" if participants failed to achieve pain freedom within 2 hours post dose. In this outcome measure, number of participants were reported according to physicians' responses. Participant who failed to achieve pain freedom at 2 hours post dose on more than half of the occasion were reported in this outcome measure.
Time Frame: 2 hours post dose (from the data collected retrospectively)
Population: Analysis population included all participants who met eligibility criteria was included in this study. Here, "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 86 | 384
Participants
  Yes | 23 | 167
  No | 63 | 217

2. Primary Outcome: Number of Participants Who Reported Migraine Pain Freedom (Success) Within 2 Hours Post Dose (Participants Perspective)
Description: Number of participants who reported migraine pain freedom within 2 hours post dosing in 0 out of every 5 attacks, 1 out of every 5 attacks, 2 out of every 5 attacks, 3 out of every 5 attacks, 4 out of every 5 attacks, or 5 out of every 5 attacks were recorded. Success was defined as responses to '4 out of every 5 attacks' or '5 out of every 5 attacks' combined. In this outcome measure, number of participants with 'success' were reported as per participants' responses. Participant who reported migraine pain freedom (success) at 2 hours post dose on more than half of occasion were reported in this outcome measure.
Time Frame: 2 hours post dose (from the data collected retrospectively)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 29 | 106
Participants | 22 | 67

3. Primary Outcome: Number of Participants Classified Based on Satisfaction With Current Acute Treatment (Physician Perspective)
Description: Physicians' satisfaction with current acute treatment for migraine was recorded and classified as extremely satisfied, satisfied, slightly satisfied, neither satisfied nor dissatisfied, slightly dissatisfied, dissatisfied and extremely dissatisfied. In this outcome measure number of participants were reported per each category according to physicians' responses.
Time Frame: Over the last 3 months prior completing the survey
Population: Analysis population included all participants who met eligibility criteria was included in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 91 | 437
Participants
  Extremely satisfied | 55 | 103
  Satisfied | 31 | 276
  Slightly satisfied | 2 | 33
  Neither satisfied nor dissatisfied | 0 | 12
  Slightly dissatisfied | 2 | 10
  Dissatisfied | 1 | 2
  Extremely dissatisfied | 0 | 1

4. Primary Outcome: Number of Participants Classified Based on Reasons for Lack of Satisfaction With Current Acute Treatment (Physician Perspective)
Description: Physicians' reported reasons for lack of satisfaction with current acute treatment. In this outcome measure number of participants were reported per each reason according to physicians' responses. There could be more than 1 reason for lack of satisfaction per participant.
Time Frame: Over the last 3 months prior completing the survey
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 5 | 58
Participants
  Lack of efficacy | 3 | 26
  Slow onset of action | 0 | 13
  Efficacy diminished over time | 0 | 17
  Number of side effects experienced | 0 | 8
  Severity of side effects experienced | 0 | 1
  Mode of administration | 0 | 2
  The number of prescribed acute treatments | 0 | 2
  The treatment is costly for the participant | 2 | 1
  Other | 1 | 7

5. Primary Outcome: Number of Participants Classified Based on Satisfaction With Current Acute Treatment (Participants Perspective)
Description: Participants' satisfaction with current acute treatment for migraine was recorded and classified as extremely satisfied, satisfied, slightly satisfied, neither satisfied nor dissatisfied, slightly dissatisfied, dissatisfied and extremely dissatisfied. In this outcome measure number of participants were reported per each category according to participants' responses.
Time Frame: Over the last 3 months prior completing the survey
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 29 | 103
Participants
  Extremely satisfied | 17 | 23
  Satisfied | 11 | 57
  Slightly satisfied | 0 | 11
  Neither satisfied nor dissatisfied | 1 | 5
  Slightly dissatisfied | 0 | 5
  Dissatisfied | 0 | 1
  Extremely dissatisfied | 0 | 1

6. Primary Outcome: Number of Participants Classified Based on Reasons for Lack of Satisfaction With Current Acute Treatment (Participants Perspective)
Description: Participants' reported reasons for lack of satisfaction with current acute treatment. In this outcome measure, number of participants were reported per each reason according to participants' responses. There could be more than 1 reason for lack of satisfaction per participant.
Time Frame: Over the last 3 months prior completing the survey
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 1 | 11
Participants
  It only reduces my migraine pain by half | 0 | 3
  It reduces my migraine pain by less than half | 0 | 1
  It does not work quickly enough | 1 | 5
  It does not work as well as it used to | 0 | 5
  The number of side effects I experience | 0 | 1
  The severity of the side effects I experience | 0 | 1
  I am not happy with the way I have to take it | 0 | 2
  I find it difficult to know when to take it | 1 | 3
  I have too many different acute treatments to take | 0 | 1
  I worry about becoming dependent on it | 0 | 1
  It costs me too much money | 0 | 1
  Other | 0 | 3

7. Primary Outcome: Number of Participants Willing to Continue Use of Acute Treatment (Participants Perspective)
Description: Participants responded about their willingness to continue use of acute treatment and responses were classified as definitely yes, probably yes, do not know, probably not, definitely not. Willingness to continue was defined as responses to: 'Definitely yes' or 'Probably yes' combined. Unwillingness to continue was defined as responses to 'Probably not' and 'Definitely not' combined. In this outcome measure number of participants were reported according to participants' responses.
Time Frame: Over the last 3 months prior completing the survey
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 29 | 94
Participants
  Willing to continue | 28 | 92
  Unwilling to continue | 1 | 2

8. Primary Outcome: Number of Participants Classified According to Responses Per Item of Migraine Treatment Optimization Questionnaire (mTOQ6)
Description: mTOQ6 was participants reported questionnaire and participants had to respond on following 6 items: 1) "Are you able to quickly return to your normal activities (i.e., work, family, leisure, social activities) after taking your migraine medication?"; 2) "After taking your migraine medication, are you pain free within 2 hours for most attacks?"; 3) "Does one dose of your migraine medication usually relieve your headache and keep it away for at least 24 hours?"; 4) "Is your migraine medication well tolerated?"; 5) "Are you comfortable enough with your migraine medication to be able to plan your daily activities?"; and 6) "After taking your migraine medication, do you feel in control of your migraines enough so that you feel there will be no disruption to your daily activities?". Each item had following responses: never, rarely, less than half the time and half the time or more.
Time Frame: Over the last 3 months prior completing the survey
Population: Analysis population included all participants who met eligibility criteria was included in this study. Here, "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure and "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 30 | 109
Participants
  Item 1: number analyzed (Participants) | 30 | 108
  Item 1: Never | 1 | 1
  Item 1: Rarely | 1 | 7
  Item 1: Less than half the time | 1 | 14
  Item 1: Half the time or more | 27 | 86
  Item 2: Never | 0 | 2
  Item 2: Rarely | 2 | 8
  Item 2: Less than half the time | 1 | 15
  Item 2: Half the time or more | 27 | 84
  Item 3: number analyzed (Participants) | 30 | 108
  Item 3: Never | 0 | 2
  Item 3: Rarely | 1 | 6
  Item 3: Less than half the time | 2 | 14
  Item 3: Half the time or more | 27 | 86
  Item 4: number analyzed (Participants) | 30 | 106
  Item 4: Never | 0 | 0
  Item 4: Rarely | 1 | 7
  Item 4: Less than half the time | 0 | 11
  Item 4: Half the time or more | 29 | 88
  Item 5: number analyzed (Participants) | 30 | 108
  Item 5: Never | 0 | 1
  Item 5: Rarely | 2 | 10
  Item 5: Less than half the time | 1 | 14
  Item 5: Half the time or more | 27 | 83
  Item 6: number analyzed (Participants) | 30 | 106
  Item 6: Never | 0 | 2
  Item 6: Rarely | 2 | 5
  Item 6: Less than half the time | 2 | 17
  Item 6: Half the time or more | 26 | 82

9. Primary Outcome: Number of Participants Classified Based on Timing They Took Acute Prescription Treatment
Description: In this outcome measure number of participants were classified based on timing/when they took acute treatment as follows: 1) before any sign of a migraine attack, but in anticipation of one starting; 2) at the first sign of a migraine attack (before the pain started); 3) when the pain started; 4) after the pain had started and participant had an idea of pain's severity.
Time Frame: Over the last 3 months prior completing the survey
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 29 | 104
Participants
  Before any sign of a migraine attack, but in anticipation of one starting | 3 | 10
  At the first sign of a migraine attack (before the pain started) | 21 | 76
  When the pain started | 4 | 15
  After the pain has started and participant had an idea of how severe it was | 1 | 3

10. Primary Outcome: Mean of Number of Days Per Month Participants Took Acute Prescription Treatment
Description: In this outcome measure mean of number of days per month participants took acute prescription treatment were recorded.
Time Frame: Over the last 3 months prior completing the survey
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days per month
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 29 | 108
Days per month | 3.29 (1.71) | 4.04 (4.82)

ADVERSE EVENTS:
Time Frame: Not applicable as adverse events were not collected for the study
Description: Due to non-interventional nature of study, the minimum criteria for reporting an adverse event (i.e., identifiable participant, identifiable reporter, a suspect product, and event) were not met, hence adverse events were not collected and reported.
Arm/Group | Rimegepant | Triptans
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT06412965/Prot_SAP_000.pdf